CLINICAL TRIAL: NCT05544006
Title: Artificial Intelligence-Based Disease Management in the Vulnerable Period of Heart Failure, An Observational Study to Evaluate Patient Speech and Voice in the Vulnerable Phase of Heart Failure
Brief Title: Artificial Intelligence-Based Disease Management in the Vulnerable Period of Heart Failure
Acronym: AIDMy-HF
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Albert Saglik Hizmetleri ve Ticaret A.S. (Industry)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Sponsor
Other Study IDs: 101052022
Record Dates: First submitted 2022-09-11; First posted 2022-09-16 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
Keywords: heart failure; vocal biomarker
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active study group: Active study group with self monitoring reminders in 3,7,14,28th days after discharge
- Usual care group: Usual care group with self monitoring recommendations at discharge

SUMMARY:
The study aims to evaluate the effect of AI-based discharge training after acute decompensation of heart failure on the patient's quality of life and to examine the relationship between changes in voice and speech characteristics of patients and changes in hospitalization, discharge, and early post-discharge clinical status.

DETAILED DESCRIPTION:
Heart failure (HF) is a progressive disease with a fluctuating course. From time to time, patients' symptoms and signs worsen enough to require hospitalization, and hospitalization occurs with acute decompensated HF. Acute HF decompensations are periods that worsen the prognosis of the patient. On the other hand, patients discharged after an acute decompensation have the highest risk during the first months after discharge. Patients get trained about lifestyle changes and medication management during the discharge period. Recent guidelines suggest that patients in the early post-discharge period be called for virtual/telephone or face-to-face control visits at short intervals(3rd, 7th, 14th, and 28th days ), then at 3-6 monthly intervals according to NYHA class.

In traditional cardiovascular practice, patients are called for outpatient control visit in the first month after discharge. However, the processes after the pandemic kept patients away from visiting the hospital at the frequency recommended in the American and European guidelines and caused them to stay at home not even following their routine visit schedules. Moreover, the risks and benefits of virtual visits in terms of patient prognosis are not well established.

This study aims to investigate relationships between routinely recorded findings, symptoms, and vocal biomarkers of heart failure patients in the hospitalization and in the post-discharge period and to investigate the effect of post-discharge education on patient-reported outcomes and re-hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation due to heart failure decompensation
* Having a smartphone with internet access
* Willingness to participate in the study
* NYHA 2-4 symptoms

Exclusion Criteria:

* Diagnosis of active malignancy
* Pregnancy
* Vision and hearing problems
* Moderate to severe cognitive impairment
* Dementia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients admitted to the Cardiology Department due to heart failure decompensation and signed a written consent will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-02 (Estimated)

PRIMARY OUTCOMES:
Heart failure-related hospitalizations | At baseline, Four weeks after discharge, Three months after discharge
  The effect of acquired intermittent digital data including vocal biomarkers along with standardized discharge education on the HF-related hospitalization
Change from baseline in health-related quality of life | At baseline, Four weeks after discharge, Three months after discharge
  The effect of acquired intermittent digital data including vocal biomarkers along with standardized discharge education on the patient's quality of life. SF-12(Short Form-12) will be used to evaluate the effect

SECONDARY OUTCOMES:
Patient-reported outcomes | At baseline, Four weeks after discharge, Three months after discharge
  Multivariate logistic regression models of digital and vocal properties optimized for sensitivity to predict patient-reported outcomes, including dyspnea level (ranging from 1 to 4), edema(0 to +3) and HF-related hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Research and Application Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Degertekin M, Erol C, Ergene O, Tokgozoglu L, Aksoy M, Erol MK, Eren M, Sahin M, Eroglu E, Mutlu B, Kozan O. [Heart failure prevalence and predictors in Turkey: HAPPY study]. Turk Kardiyol Dern Ars. 2012 Jun;40(4):298-308. doi: 10.5543/tkda.2012.65031. Turkish. PMID 22951845
- [Background] Yilmaz MB, Celik A, Cavusoglu Y, Bekar L, Onrat E, Eren M, Kutlu M, Yalta K, Temizhan A, Kilicaslan B, Gungor H, Acikel M, Demir M, Akdemir R, Zoghi M, Tokgozoglu L. [Snapshot evaluation of heart failure in Turkey: Baseline characteristics of SELFIE-TR]. Turk Kardiyol Dern Ars. 2019 Apr;47(3):198-206. doi: 10.5543/tkda.2019.66877. Turkish. PMID 30982817